CLINICAL TRIAL: NCT06377891
Title: The Effect of Emotional Resilience Training on Fear of Birth and Depression in Primiparous Pregnant Women: Randomized Controlled Study
Brief Title: The Effect of Emotional Resilience Training on Fear of Birth and Depression in Primiparous Pregnant Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Elif Odabası Aktas, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TDK-2024-13563
Record Dates: First submitted 2024-04-15; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Fear of Childbirth; Depression
Keywords: Resilience; Pregnant; Primiparous; Fear of Childbirth; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Resilience Group (Experimental): Providing emotional resilience training to the experimental group.
  Interventions: Other: Emotional Resilience training
- Control group (No Intervention): There will be no intervention in the control group.

INTERVENTIONS:
Other: Emotional Resilience training — Primiparous pregnant women in the experimental group will be given emotional resilience training in the last trimester.
  Arms: Emotional Resilience Group

SUMMARY:
Although birth has a great place in a woman's life, factors such as the woman's education level, personal experiences, social support status, whether the pregnancy is planned or not, the family's attitude towards pregnancy, and socioeconomic status increase the burden of pregnancy and can create a stressful situation for the woman. While the pain that may be experienced during birth, thoughts about the baby's health and postpartum baby care further increase this fear, primiparous women who will give birth for the first time experience many emotions that they cannot define and cannot predict the situations they will encounter during birth. The most important situation that will cause pain during birth is fear. So much so that fear of birth may cause women to avoid pregnancy and increase optional abortions.In particular, fear of birth may increase cesarean delivery rates and also lead to negative maternal outcomes such as poor mental health after birth. Fear experienced during the antenatal period can lead to difficult births, mother-baby attachment problems, and depression. While fear of birth causes depression and anxiety disorders in the postpartum period, it is stated that depression experienced during pregnancy may increase the fear of birth, or fear of birth may be a hidden symptom of depression. It is noted that emotional regulation skills and resilience in pregnant women can be effective strategies in minimizing and managing fear, anxiety, stress, and anxiety. Emotional resilience is defined as the style of coping with stress, the ability to repair oneself, the ability to recover from adverse events quickly, and the state of adapting to a new environment. In particular, individuals with high emotional resilience can protect their physical and mental health and increase their life satisfaction by reducing the negative consequences they experience. With the emotional resilience training given during pregnancy, pregnant women's stress, fear, and anxiety will be reduced, and they will be able to cope better with the difficulties they experience. This research will be conducted to examine the effect of emotional resilience training given to primiparous pregnant women on fear of childbirth and depression.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Volunteering to participate in the research,
* 32-34. Being at the gestational age,
* Knowing Turkish,
* Being at least a primary school graduate,
* Having a single and healthy fetus,
* Having a WBDRS-A score of 38 and above,
* Being at least a primary school graduate.
* Depression score above 12/13,

Exclusion Criteria:

* Pregnant women with any risky pregnancy history (Preeclampsia, placenta previa, gestational diabetes mellitus, oligohydramnios and polyhydroamnios, etc.),
* Those who do not attend at least one of the sessions of the training program,
* Chronic and/or psychiatric health Pregnant women with problems (based on self-report and clinical diagnosis status) will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-04-16 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The effect of emotional resilience on fear of birth and depression in primiparous pregnant women. | 32-34 gestational weeks - 4 follow-ups until the 6th week postpartum
  To make the effect of emotional resilience training given to primiparous pregnant women on fear of birth and depression during pregnancy and after birth visible with WIJMA-A and WIJMA-B fear of birth scale (Low (score ≤ 37), moderate (38-65), severe (66-84) and clinical fear of birth (≥ 85)) and Edinburgh depression scale (The cut-off point was calculated as 12/13, and women whose total scale score is more than the cut-off point are considered to be in the risk group)

CONTACTS AND LOCATIONS:
Locations (1):
- Bayburt State Hospital, Bayburt, Turkey (Türkiye)